CLINICAL TRIAL: NCT03328338
Title: Mitochondrial Function in Transthyretin Amyloidosis : the MIT-AMYLOSE Study.
Brief Title: Mitochondrial Function in Transthyretin Amyloidosis
Acronym: MIT-Amylose
Status: Terminated | Type: Observational
Why Stopped: Mitochondrial respiration measurement technique faulty
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Other Study IDs: 16/E/17
Record Dates: First submitted 2017-10-28; First posted 2017-11-01 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Cardiac Amyloidosis
Keywords: Mitochondria; Oxidative phosphorylation (mitochondrial respiration); Subcutaneous abdominal adipose tissue; Heart.
MeSH Terms: conditions — Amyloid Neuropathies, Familial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hereditary (familial) amyloidosis arising from the misfolding of a mutated or variant transthyretin, is the most frequent form of amyloid cardiomyopathy in the Caribbean basin. Affected organs invariably harbor extracellular amyloid deposits in the myocardium. Circulating or pre-fibrillar amyloidogenic proteins are implicated in the disruption of cell function. The investigators aim is to demonstrate that transthyretin mediated amyloid disease alter the mitochondrial function of cardiac cells.

DETAILED DESCRIPTION:
Systemic amyloidosis are a family of diseases induced by misfolded and/or misassembled proteins. Extracellular deposits of these proteins disrupt vital organ function. Two types of amyloid commonly infiltrate the heart: immunoglobulin light-chain amyloid and transthyretin (TTR) amyloid. Among the TTR variants that predominantly target the heart, the valine to isoleucine substitution at position 122 (V122I or Ile122) is the most common. This TTR variant is responsible for the most frequent form of amyloid cardiomyopathy in the Caribbean basin. Increasingly study data supports a central role for circulating or pre-fibrillar amyloidogenic proteins in the disruption of cardiac function in TTR mediated amyloid disease. In vivo exposure of cultured cardiomyocytes to pre-fibrillar an amyloidogenic proteins stimulate the production of reactive oxygen species and disrupts calcium fluxes. (Recent studies indicate that pre-fibrillar amyloidogenic proteins may also induce apoptosis through the mitochondrial pathway, eventually leading to cardiac cell injury). Hence, growing evidence suggests that end-organ damage by pre-fibrillar TTR amyloid may be related to mitochondrial dysfunction. Diagnosis of cardiac amyloidosis can be based on invasive heart biopsies or a non-invasive approach including identification of amyloid tissue deposits from abdominal fat biopsies. The investigators aim is to demonstrate that transthyretin mediated amyloid disease alters the mitochondrial function of subcutaneous abdominal adipocytes.

The investigators objective is to study mitochondrial respiration assessed by oxygraphy in fragments of subcutaneous abdominal fat biopsies performed for diagnosis of TTR amyloidosis. Mitochondrial respiration will be evaluated in the absence and in the presence of ADP.

Follow the evaluation of mitochondrial respiration. So, no patient follow-up will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Have a parietal thickness measuring more than 15 mm on the echocardiography or have structural and echogenicity abnormalities characteristic of cardiac amyloidosis,
* Live in Martinique,
* Accept the use of the residues coming from biopsies of the subcutaneous abdominal adipose tissue performed during the medical care.

Exclusion Criteria:

* Be under 18 years old,
* Have a contraindication to subcutaneous biopsy,
* Be allergic to local anesthetics,
* Pregnant or nursing woman,
* Have a cardiovascular disease suggesting a secondary cardiac disease, such as documented severe hypertension, valvular stenosis, or a known familial cardiomyopathy,
* Be major under guardianship / curatorship or deprived of liberty,
* Not be able to answer to a simple administrative questionnaire or to give freely its non-opposition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The selection of patients is done during the amyloidosis consultation of the cardiology department.
  Patients are referred to this consultation following the discovery of characteristic abnormalities during echocardiography.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-29 (Actual)

PRIMARY OUTCOMES:
Oxygen consumption measure in subcutaneous abdominal fat biopsies | Three months
  The mitochondrial respiration of the cells is measured by polarography with a "Clark" type oxygen electrode. The Clark electrode consists of a platinium cathode and a silver anode. When a potential difference of -0.6 volts is applied, the platinium electrode is negatively charged with respect to that of silver and each oxygen molecule dissolved in the medium diffuses through the gas-permeable Teflon membrane, and is reduced at the cathode according to the following reaction: O 2 + 4H + + 4e → 2H 2 O. The current thus generated is proportional to the concentration of dissolved oxygen. The oxygen saturation constant (406 nmol / ml) makes it possible to convert these results into oxygen consumption / minute.

SECONDARY OUTCOMES:
Rates of oxygen consumption | Three months
  Rates of oxygen consumption (expressed as pmol O2.s-1.mg of fat tissue) will be recorded in-vivo in different conditions, which include routine respiration and after ADP addition. Carbonyl cyanide-4-(trifluoromethoxy) phenylhydrazone (FCCP), tetra methyl-p-phenylenediaminedihydrochloride (TMPD)-ascorbate and oligomycin will be tested in vitro to monitor uncoupled respiration, cytochrome c oxidase activity and leak state respiration by inhibition of ATP synthase, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyn INAMO, MD-PhD, Principal Investigator — CHU de Martinique
Locations (1):
- CHU de Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD, all IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After the main publication of the results, for not limited time.
Access Criteria: The conditions for the transfer of all or part of the database of the research are decided by the investigator coordinator / sponsor of the research and are the subject of a written contract.

REFERENCES:
- [Background] Inamo J, Daigre JL, Boissin JL, Kangambega P, Larifla L, Chevallier H, Balkau B, Smadja D, Atallah A. High blood pressure and obesity: disparities among four French Overseas Territories. J Hypertens. 2011 Aug;29(8):1494-501. doi: 10.1097/HJH.0b013e328348fd95. PMID 21720269
- [Result] Oliveira Da Silva L, Fabre J, Monfort A, Villeret J, Citony I, Cohen-Tenoudji P, Lebbadi M, Martin D, Molinie V, Inamo J. 'Green Apple' Heart Failure. West Indian Med J. 2014 Jul 3;63(6):673-5. doi: 10.7727/wimj.2013.255. Epub 2014 Jun 25. PMID 25803389
- [Result] Parent F, Bachir D, Inamo J, Lionnet F, Driss F, Loko G, Habibi A, Bennani S, Savale L, Adnot S, Maitre B, Yaici A, Hajji L, O'Callaghan DS, Clerson P, Girot R, Galacteros F, Simonneau G. A hemodynamic study of pulmonary hypertension in sickle cell disease. N Engl J Med. 2011 Jul 7;365(1):44-53. doi: 10.1056/NEJMoa1005565. PMID 21732836
- [Result] Montaigne D, Marechal X, Coisne A, Debry N, Modine T, Fayad G, Potelle C, El Arid JM, Mouton S, Sebti Y, Duez H, Preau S, Remy-Jouet I, Zerimech F, Koussa M, Richard V, Neviere R, Edme JL, Lefebvre P, Staels B. Myocardial contractile dysfunction is associated with impaired mitochondrial function and dynamics in type 2 diabetic but not in obese patients. Circulation. 2014 Aug 12;130(7):554-64. doi: 10.1161/CIRCULATIONAHA.113.008476. Epub 2014 Jun 13. PMID 24928681
- [Result] Montaigne D, Marechal X, Lefebvre P, Modine T, Fayad G, Dehondt H, Hurt C, Coisne A, Koussa M, Remy-Jouet I, Zerimech F, Boulanger E, Lacroix D, Staels B, Neviere R. Mitochondrial dysfunction as an arrhythmogenic substrate: a translational proof-of-concept study in patients with metabolic syndrome in whom post-operative atrial fibrillation develops. J Am Coll Cardiol. 2013 Oct 15;62(16):1466-73. doi: 10.1016/j.jacc.2013.03.061. Epub 2013 May 1. PMID 23644086
- [Result] Preau S, Montaigne D, Modine T, Fayad G, Koussa M, Tardivel M, Durocher A, Saulnier F, Marechal X, Neviere R. Macrophage migration inhibitory factor induces contractile and mitochondria dysfunction by altering cytoskeleton network in the human heart. Crit Care Med. 2013 Jul;41(7):e125-33. doi: 10.1097/CCM.0b013e31827c0d8c. PMID 23478658